CLINICAL TRIAL: NCT05621707
Title: A Phase 2 Trial of Concurrent Chemoradiotherapy Following Immunotherapy Plus Chemotherapy for Patients With Locally-advanced Esophageal Squamous Cell Cancer
Brief Title: Chemoradiotherapy Following Immunotherapy Plus Chemotherapy for Locally-advanced Esophageal Squamous Cell Cancer (RICE)
Acronym: RICE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: drjunliu
Record Dates: First submitted 2022-11-05; First posted 2022-11-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinomas; Concurrent Chemoradiotherapy; Immunotherapy; Chemotherapy
Keywords: esophageal cancer; chemoradiotherapy; immunotherapy; chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Induction Therapy: Two cycles of induction chemotherapy (nab-paclitaxel 200 mg/m², day 1; carboplatin AUC 5, day 1) combined with a PD-1 inhibitor (200 mg, day 1) every 3 weeks.
  Concurrent Therapy: Followed by concurrent chemoradiotherapy (CCRT).
  Maintenance Therapy: Patients without progressive disease (PD) will receive maintenance immunotherapy with a PD-1 inhibitor (200 mg every 3 weeks) for up to 1 year.
  Interventions: Drug: chemotherapy combined with PD-1 inhibitors

INTERVENTIONS:
Drug: chemotherapy combined with PD-1 inhibitors — Induction chemotherapy combined with PD-1 inhibitors followed with standard concurrent chemoradiotherapy

SUMMARY:
This is an investigator-initiated, single-arm, exploratory clinical study.The study population consisted of non-operative Locally Advanced Esophageal Cancer . The purpose of this study was to evaluate the efficacy and safety of Concurrent Chemoradiotherapy Following Immunotherapy Plus Chemotherapy for Patients With Locally-advanced Esophageal Squamous Cell Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of screening.
2. Histologically confirmed squamous cell carcinoma;
3. Locally-advanced ,medical inoperability, technical irresectability, or patient refusal to surgery;
4. Eastern Cooperative Oncology Group (ECOG) performance status:0-2;
5. Able to eat a semi-liquid diet;
6. Less than 20% weight loss within 6 months;
7. Adequate hepatic function, renal function, hematologic function and coagulation function;
8. Documented informed consent.

Exclusion Criteria:

1. Distant metastasis;
2. Known malignancy diagnosed or require active treatment in the last 5 years, except for cancers that can be cured by surgery including cervical cancer in situ, basal or squamous cell skin cancer, breast ductal carcinoma in situ, localized prostate cancer;
3. Prior thoracic irradiation, chemotherapy, or lobectomy
4. Known diseases or conditions that are contraindicated for radiotherapy or surgery;
5. Allergy to the research medications;
6. Pregnant women or women preparing for pregnancy;
7. Diagnosis of autoimmune disease or history of chronic autoimmune disease
8. Absence of informed consent because of psychological, family, social and other factors;
9. Patients with comorbidities (chronic pulmonary disease, poorly controlled hypertension, unstable angina, myocardial infarction within 6 months, unstable mental disorders requiring therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate | 2 years after last patient enrolled
  Overall survival rate is defined as the percentage of participants who are alive up to 2 years from enrollment

SECONDARY OUTCOMES:
progression-free Survival (PFS) | 2 years after last patient enrolled
  Progression-free survival is defined as the time between date of enrollment and first date of recurrence or death, whichever occurs first.Recurrence is defined as the appearance of one or more new lesions, which can be local, regional, or distant in location from the primary tumor site ( assessed by imaging or pathology). All deaths without prior recurrence are considered as PFS events.
Treatment related complications | During the procedure
  complications after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China